CLINICAL TRIAL: NCT05585736
Title: Effect of Cycloplegia on the Refractive Status of Egyptian Children
Brief Title: Cycloplegia and Refractive Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ehab tharwat, Principal Investigator, Al-Azhar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Cycloplegia
Record Dates: First submitted 2022-09-17; First posted 2022-10-19 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Cycloplegia
MeSH Terms: interventions — Mydriatics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cycloplegic refraction (Other): All refractions were measured before and after cycloplegic addition to the eye.
  Interventions: Drug: Cycloplegics

INTERVENTIONS:
Drug: Cycloplegics — they are drugs that paralyze the ciliary muscles and cause relaxation of accommodation.

SUMMARY:
Myopia is a public health problem, affecting the general population worldwide. The common modalities for correcting myopia include spectacles, contact lenses, and surgical procedures. Cycloplegic refraction is considered the gold standard for measuring refractive errors, especially in children. It has been well-established that generally myopia could be overestimated and hyperopia be underestimated if refraction was performed without cycloplegia.

ELIGIBILITY:
Inclusion Criteria:

* Myopia or Hyperopia or compound myopic astigmatism.
* Normal intra ocular pressure (IOP≤21 mmHg.
* Age > 2 years and < 10 years

Exclusion Criteria:

* Unwilling to participate in the study.
* Previous ocular surgery
* Any diagnosed ocular disease
* History of ocular trauma
* Irregular astigmatism on corneal topography.

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 388 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Sphere of the eye | Baseline
  It means that the correction for nearsightedness or farsightedness is spherical, equal in all meridians of the eye. This indicates the amount of lens power, measured in diopters (D), prescribed to correct nearsightedness or farsightedness. If the number appearing under this heading has a minus sign (-), you are nearsighted; if the number has a plus sign (+) or is not preceded by a plus sign or a minus sign, you are farsighted. It is measured by Auto-refractor
Sphere of the eye | Immediate after 30 minutes of cycloplegic addition
  It means that the correction for nearsightedness or farsightedness is spherical, equal in all meridians of the eye. This indicates the amount of lens power, measured in diopters (D), prescribed to correct nearsightedness or farsightedness. If the number appearing under this heading has a minus sign (-), you are nearsighted; if the number has a plus sign (+) or is not preceded by a plus sign or a minus sign, you are farsighted. It is measured by Auto-refractor
cylinder of the eye | Baseline
  This indicates the amount of lens power for astigmatism and represents the difference in the greatest and weakest powers of the eye, usually separated by 90 degrees. If nothing appears in this column, either you have no astigmatism, or your astigmatism is so slight that it is not necessary to correct it with your eyeglass lenses. The number in the cylinder column may be preceded with a minus sign (for the correction of nearsighted astigmatism) or a plus sign (for farsighted astigmatism). Cylinder power always follows sphere power in an eyeglass prescription. It is measured by Autorefractor.
cylinder | Immediate after 30 minutes after cycloplegia
  This indicates the amount of lens power for astigmatism and represents the difference in the greatest and weakest powers of the eye, usually separated by 90 degrees. If nothing appears in this column, either you have no astigmatism, or your astigmatism is so slight that it is not necessary to correct it with your eyeglass lenses. The number in the cylinder column may be preceded with a minus sign (for the correction of nearsighted astigmatism) or a plus sign (for farsighted astigmatism). Cylinder power always follows sphere power in an eyeglass prescription. It is measured by Autorefractor

CONTACTS AND LOCATIONS:
Locations (1):
- Ehab tharwat, Damietta, New Damietta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided